CLINICAL TRIAL: NCT02428946
Title: Bromocriptine and Insulin Sensitivity in Lean and Obese Subjects
Brief Title: Bromocriptine and Insulin Sensitivity
Acronym: BIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, F Holleman, Dr. MD., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: NL49417.018.14 METC 2014/147
Record Dates: First submitted 2014-10-17; First posted 2015-04-29 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Insulin Sensitivity
Keywords: Insulin Sensitivity; obesity; dopamine
MeSH Terms: conditions — Insulin Resistance; Obesity | interventions — Bromocriptine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morning bromocriptine (Active Comparator): Bromocriptine is taken in the morning
  Interventions: Drug: Bromocriptine
- Evening bromocriptine (Active Comparator): Bromocriptine is taken in te evening
  Interventions: Drug: Bromocriptine

INTERVENTIONS:
Drug: Bromocriptine — Investigating the randomized order for timing of bromocriptine administration
  Other Names: Parlodel

SUMMARY:
In this study the investigators will examine the effect of dopamine (bromocriptine) on insulin sensitivity in lean and obese subjects. Furthermore, the investigators will examine whether the timing of bromocriptine administration has influence on insulin sensitivity.

To do so, the investigators will include lean and obese subjects who will use 2 times 2 weeks bromocriptine. In randomized order, they will use it in the morning or in the evening.

The investigators will examine insulin sensitivity by performing a 7-point oral glucose tolerance test.

Furthermore, the investigators will examine energy expenditure and subjects will keep track of their eating behaviour in the 3 days before each study visit.

DETAILED DESCRIPTION:
Bromocriptine, a dopamine 2 receptor agonist, has recently been approved in the treatment of type 2 diabetes mellitus(DM2). Bromocriptine causes a significant improvement of fasting plasma glucose and Hba1C values. The exact mechanism of action of bromocriptine is still unknown.

Earlier, the investigators performed a study to show the effects of bromocriptine on brown adipose tissue (BAT) activity (the DEBAT study (Medisch Etische Toetsingscommissie) METC nr 2013_107). Namely, BAT, known for its capacity to dissipate excess energy, might have been involved in this process as stimulation by the sympathetic nervous system is the principal driving force in controlling BAT activity. However, the investigators have shown that bromocriptine did not influence BAT activity or energy expenditure in healthy, lean subjects.

The investigators did found an effect of bromocriptine on insulin sensitivity unexpectedly, subjects became significantly less insulin sensitive after bromocriptine use.

Circadian neuroendocrine rhythms, especially the dopaminergic and serotonergic neurotransmitter activity, play a pivotal role in the development of seasonal and non-seasonal changes in body fat stores and insulin sensitivity. Therefore, the timing of bromocriptine administration might be of great importance in changes in insulin sensitivity. Indeed, in the treatment for DM2, a bromocriptine quick release variant is given in the morning. In the former study the investigators instructed the subjects to use the bromocriptine in the evening in combination with the evening meal. The investigators decided to do so because bromocriptine had to be taken in combination with food. The investigators wanted a high level of dopamine just before the 18F-Fludeoxyglucose(18F-FDG) positron emission tomography (PET) computed tomography (CT) scan to get a maximum effect of dopamine on BAT. But the subjects had to be fasted for the OGTT and 18F-FDG-PET-CT scan. Therefore, the investigators decided to give the (long-acting) bromocriptine in the evening.

Also, the effect of bromocriptine might be different in lean or obese subjects. Obesity is associated with an increased sympathetic tonus. Therefore, the baseline condition is different in lean or obese subjects which may cause different effects of bromocriptine treatment.

In this study the investigators aim to investigate whether the timing (e.g. morning or evening) of bromocriptine administration (1,25mg/day during the first week and 2,50mg/day during the second week) has different effects on insulin sensitivity in both lean and obese males.

At visit 1: Informed consent, medical history, vital signs and laboratory measurements will be obtained. The investigators will also perform an oral glucose tolerance test (OGTT), and an energy expenditure(EE) measurement after 60 minutes bed rest.

After visit 1: subjects will start using bromocriptine (1,25mg/day during the first week and 2,50mg/day during the second week) randomization to timing: in the morning or evening.

Visit 2: EE after 60 minutes rest. OGTT. 2 weeks washout period Visit 3: EE after 60 minutes rest. OGTT. After visit 3: start using bromocriptine (1,25mg/day during the first week and 2,50mg/day during the second week) at other time point.

Visit 4: EE after 60 minutes rest. OGTT.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian origin
* Subjects should be able and willing to give informed consent
* BMI range of 19-23 kg/m2 or BMI> 27 kg/2

Exclusion Criteria:

* Renal failure (creatinine>135mmol/l)
* Liver failure (ASAT/ALAT > 3 times higher than the normal upper value)
* Daily use of prescription medication
* Known hypersensitivity to bromocriptine.
* Uncontrolled hypertension
* Known history of coronary artery disease or valvulopathy
* History of severe psychiatric disorders.
* Prolactin-releasing pituitary tumor (prolactinoma).

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Timing of administration of bromocriptine | 6 weeks
  To determine whether there is a beneficial effect on insulin sensitivity when bromocriptine is given in the morning, as compared to bromocriptine in the evening in Caucasian, lean and obese males

SECONDARY OUTCOMES:
Difference in insulin sensitivity between lean and obese males before and after the use of bromocriptin | 6 weeks
  To determine whether there are differential effects of bromocriptine treatment on insulin sensitivity in obese or lean healthy, Caucasian males
Difference in energy expenditure in lean and obese before and after the use of bromocriptin | 6 weeks
  To determine whether the difference in timing of bromocriptine influences energy expenditure during thermoneutral conditions in Caucasian, lean and obese males

CONTACTS AND LOCATIONS:
Overall Officials: Frits Holleman, Dr. MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands